CLINICAL TRIAL: NCT04475913
Title: In a Post -Covid-19 World, What is the Clinical Influence of Digital vs Analog Impression in Cases of All-on-4 - Prosthesis ?
Brief Title: Digital vs Analog Impression in Cases of All-on-4 - Prosthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October University for Modern Sciences and Arts (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5
Record Dates: First submitted 2020-07-14; First posted 2020-07-17 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2020-07

CONDITIONS: Edentulous Mouth
Keywords: impressions; analogue; digital; All-on-Four
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- (CIG Axial) (Active Comparator): received 4 axial implants and conventional impression
  Interventions: Other: DIG Axial
- (DIG Axial) (Experimental): received 4 axial implants and digital impression
  Interventions: Other: DIG Tilted; Other: CIG Axial
- CIG Tilted (Active Comparator): received two anterior axial implants and two distal tilted implants, and conventional impression
  Interventions: Other: DIG Tilted
- (DIG Tilted) (Experimental): received two anterior axial implants and two distal tilted implants, and digital impression
  Interventions: Other: DIG Axial; Other: CIG Tilted

INTERVENTIONS:
Other: DIG Axial — patients received 4 axial implants and digital impression
  Arms: (CIG Axial); (DIG Tilted)
Other: DIG Tilted — received two anterior axial implants and two distal tilted implants, and digital impression
  Arms: (DIG Axial); CIG Tilted
Other: CIG Axial — patients received 4 axial implants and conventional impression
  Arms: (DIG Axial)
Other: CIG Tilted — received two anterior axial implants and two distal tilted implants, and conventional impression
  Arms: (DIG Tilted)

SUMMARY:
Fifty six patients were randomly enrolled in the study. Participants were randomly stratified into two control groups and two test groups, from which conventional pick up and digital impressions were made respectively. Patients of group 1 (CIG Axial) and 3 (DIG Axial) received 4 axial implants whereas, group 2 patients (CIG Tilted), and group 4 (DIG Tilted) received two anterior axial implants and two distal tilted implants.

All participants received hybrid dentures. Bone loss, implant loss, maintenance of prosthesis were evaluated at 6m,12m, and 24 months follow up period.

ELIGIBILITY:
Inclusion Criteria:

* completely edentulous patients with age range from 50-65 years.
* physically and psychologically eligible participants for implants placement.
* adequate bone to receive 4 interforaminal implants.

Exclusion Criteria:

participants were excluded if

* medical conditions that precludes implants placement
* smokers
* patients suffering from any parafunctional habits

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2020-07-11 (Actual); Study Completion 2020-08-20 (Actual)

PRIMARY OUTCOMES:
implant loss | 24 months
  The implants were considered surviving if they were clinically stable and functioning without any mobility. Failure was defined removal of implants due to loss of integration, pain, implant mobility, paraesthesia, neuropathies or psychological reasons. Calculation of the estimated failure rate was performed by dividing the number of implant failures by the total exposure time of the implant. The total exposure time is the interval of time the implants could be followed for the entire observation time or up to failure of the implants that were lost during the follow-up period.

SECONDARY OUTCOMES:
crestal bone loss | 24 months
  Standardized periapical radiographs with long cone paralleling technique using film holders were used for the assessment of crestal bone loss. The loss of marginal bone relative to the implant shoulder at the mesial and distal of each implant was measured in mm and then the mean was calculated and statistically estimated. A digital intraoral imaging system was used (Digora phosphor plate reader, Soredex Tuusula, Finland). All the radiographs were scanned and then uploaded into the computer for assessing bone loss over time. The "ImageJ" software was used to take the measurements on the computer screen. Postoperative radiographs with the implants placed at the crest of the bone were compared with the 6,12 and 24 m radiographs.

OTHER OUTCOMES:
maintenance | 24 months
  During the follow-up period, prosthodontic (mechanical) complications for the four groups were registered and calculated according to the following events: number of screw loosening or screw fracture of the abutment, number of screw loosening or screw fracture of the prosthesis, number of framework fracture, fractured acrylic resin, number of prosthetic teeth fracture and loss of cover of access hole.

CONTACTS AND LOCATIONS:
Overall Officials: Dina Elawady, Principal Investigator — Lecturer
Locations (1):
- OctoberUMSA, Giza, Egypt